CLINICAL TRIAL: NCT04973696
Title: Toolkit for Optimal Recovery After Orthopedic Injury; A Multisite Feasibility Study to Prevent Persistent Pain and Disability
Brief Title: Toolkit for Optimal Recovery After Orthopedic Injury
Acronym: TOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Texas at Austin (Other); University of Kentucky (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020P000095
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Results first posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Acute Orthopedic Injury
Keywords: Mind-Body; Pain; Physical Function; Disability; Psychosocial
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Research assistants who assess outcomes and collect data after randomization, orthopedic surgeons, and statistician will be blinded.
  The study clinicians will be unblinded. The research assistant who enrolls participants and performs activities before randomization will be unblinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toolkit for Optimal Recovery after Orthopedic Injury - Active (Experimental): The Toolkit (TOR) is a 4-session, individual, live video, synchronous program developed specifically for patients with orthopedic acute injuries who are at risk for chronic pain and disability. The program teaches evidence-based mind-body skills (e.g., relaxation and mindfulness; myths about pain; activity pacing; acceptance and values based goal setting). Participants gain access to a website downloaded on their phones as an app. The website included explainer videos of skills and recordings of mindfulness and relaxation exercises. In addition, participants will receive usual care as determined by medical team.
  Interventions: Behavioral: Toolkit for Optimal Recovery after Orthopedic Injury
- Minimally Enhanced Usual Care (MEUC) - Control (Active Comparator): The MEUC is educational material, in the form of a physical hard-copy pamphlet and website downloaded as an app on their phones. In addition, participants will receive usual care as determined by medical team.
  Interventions: Other: Minimally Enhanced Usual Care (MEUC)

INTERVENTIONS:
Behavioral: Toolkit for Optimal Recovery after Orthopedic Injury — The Toolkit (TOR) is a 4-session, individual, live video, synchronous program developed specifically for patients with orthopedic acute injuries who are at risk for chronic pain and disability. The program teaches evidence-based mind-body skills (e.g., relaxation and mindfulness; myths about pain; activity pacing; acceptance and values based goal setting). Participants gain access to a website downloaded on their phones as an app. The website included explainer videos of skills and recordings of mindfulness and relaxation exercises. In addition, participants will receive usual care as determined by medical team.
  Arms: Toolkit for Optimal Recovery after Orthopedic Injury - Active
Other: Minimally Enhanced Usual Care (MEUC) — The MEUC is educational material, in the form of a physical hard-copy pamphlet and website downloaded as an app on their phones. In addition, participants will receive usual care as determined by medical team.
  Arms: Minimally Enhanced Usual Care (MEUC) - Control

SUMMARY:
This is a multi-site randomized feasibility trial of the Toolkit for Optimal Recovery after Orthopedic Injury (TOR), a mind-body program to prevent persistent pain and disability in at-risk patients with acute orthopedic injury, versus a minimally-enhanced usual care (MEUC) control. TOR is a 4-session program delivered via secure live video to patients at risk for chronic pain, 1-2 months after an orthopedic traumatic injury. The primary aim of this study is to determine whether the study methodology (i.e., implementation, randomization, procedures and assessment of outcome measures) and delivery of TOR meet a priori set benchmarks for feasibility, acceptability, and appropriateness, necessary for the success of the subsequent efficacy trial.

DETAILED DESCRIPTION:
Study Rationale:

The care of patients with acute orthopedic injuries follows an outdated biomedical model, and consists primarily of surgical interventions and pain medications, despite strong evidence for the pivotal role of psychosocial factor in transition to persistent pain and disability.

We developed the first mind-body program - The Toolkit for Optimal Recovery after orthopedic injury (TOR) - to prevent chronic pain and disability in at-risk patients with orthopedic injuries. TOR is based on the fear avoidance model and teaches skills (e.g., mindfulness and relaxation, adaptive thinking, acceptance) to help optimize recovery. Each TOR session is 45 minutes long, and there are 4 sessions delivered within a period of 4-5 weeks (TOR and control arm will be yoked for the timing of interventions).

Primary Objective The primary objective is to conduct a multi-site feasibility RCT of TOR versus MEUC control in order to determine whether the study methodology and TOR meet a priori set benchmarks necessary for the success of the subsequent efficacy trial. There are 5 primary outcomes: 1. Feasibility of recruitment (assessed by number of participants who agree to participate); 2. Appropriateness (assessed with the Credibility and Expectancy Scale); 3. Feasibility of data collection (self-report; assessed by number of participants who complete these measures at the 3 time points); 4. Treatment satisfaction (assessed with the Client Satisfaction Scale); and 5. Acceptability of TOR (adherence to sessions).

It should be noted that some of the feasibility outcomes/markers will be reported for both groups together (i.e. TOR and MEUC combined, for example the feasibility of data collection), but others were only collected and reported for the TOR group, because they were assessing the intervention specifically; the intervention was only administered in the TOR arm, and thus this outcome can only be reported for the TOR arm. Outcomes will clearly state which groups they are reported for, if results are combined, and rationale will be provided for this decision.

Hypothesis: We expect that TOR will meet all a priori set benchmarks.

Secondary Objectives:

There will be 27 secondary outcomes. Outcomes (both primary and secondary) will be reported for all sites combined, unless otherwise noted in an outcome description. Several secondary outcomes (which will be noted) will assess whether the intervention (TOR) tested in this study is feasible, acceptable, and satisfactory, from the point of view of the staff and surgeons in the orthopedic clinics (sites of recruitment for intervention participants). These feasibility secondary outcomes do not reflect the perspectives or numbers of the actual participants (180 planned) who were enrolled in the trial, but rather those of the staff and surgeons in the clinics where these participants are being treated for their orthopedic injury, and from which referrals for participation in the study came.

Study Design:

In the present study, 180 patients with acute orthopedic injuries from the Level I Trauma Centers at Massachusetts General Hospital (Boston, MA), Dell Medical School (Austin, TX), the University of Kentucky (Lexington, KY), and Vanderbilt University Medical Center (Nashville, TN) who are at risk for chronic pain and disability are planned to be enrolled. After consent and baseline assessments, participants will be randomly assigned to TOR or to a minimally enhanced usual care control (MEUC). Subjects in the TOR group undergo a 4-week session (~45 minutes each), individual, live video, synchronous mind-body intervention. The MEUC group will receive a pamphlet containing brief summarized information that reflects the intervention topics (e.g., the trajectory of pain and recovery after orthopedic illness). In addition, participants in both groups will receive usual medical care as determined by the medical team. Participants in both groups will complete assessments at baseline, after the completion of TOR, and 3 months (from baseline) later.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female outpatients in the Level 1 Trauma Center of one of the 4 sites, age 18 years or older
2. Sustained one more more acute orthopedic injuries (e.g., fracture, dislocation, rupture) approximately 1-2 months earlier (acute phase)
3. Score ≥20 on the Pain Catastrophizing Scale (PCS) or ≥40 on the Short Form Pain Anxiety Scale (PASS-20)
4. Willing to participate and comply with the requirements of the study protocol, including randomization, questionnaire completion, and potential home practice and weekly sessions.
5. No psychotropics for at least 2 weeks prior to initiation of treatment or stable for >6 weeks and willing to maintain a stable dose
6. Cleared by orthopedic surgeon for activities using the injured limb within the next 4 weeks
7. Able to meaningfully participate (e.g., English speaking and comprehension, stable living situation as determined by the medical staff at each site)
8. A score of 8/10 or more on the Short Portable Mental Status Questionnaire ONLY IF a participant is 65 or older, or if a participant's cognitive abilities are unclear to research staff

Exclusion Criteria:

1. Serious comorbidity expected to worsen in the next 3 months (e.g., malignancy)
2. Current untreated or unstable severe mental health conditions like bipolar disorder, schizophrenia, or active substance use
3. Current suicidal ideation
4. Other unmanaged serious non-orthopedic injuries that occurred alongside the orthopedic injury (i.e., TBI, ruptured internal organs, etc.)
5. Practice of meditation, or other mind body techniques that elicit the RR, for at least 45 total minutes a week each week over the last 3 months
6. Currently in litigation or under Workman's Comp
7. Surgery complications (e.g., uncontrolled infection, need for repeat surgery)
8. Self-reported pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maria Vranceanu, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The two arms for this study and participant flow are listed below. As stated in the Protocol Section, several secondary outcomes will assess whether the intervention (TOR) tested in this study is feasible, acceptable, and satisfactory, from the point of view of the clinic staff and surgeons in the orthopedic clinics that are the sites of recruitment for study participants. Since they were not actually enrolled in the study, these clinic staff and surgeons are not included in participant flow.
Groups:
- Toolkit for Optimal Recovery After Orthopedic Injury (TOR) - Active: Toolkit for Optimal Recovery after Orthopedic Injury: The Toolkit (TOR) is a 4-session, individual, live video, synchronous program developed specifically for patients with orthopedic acute injuries who are at risk for chronic pain and disability. The program teaches evidence-based mind-body skills (e.g., relaxation and mindfulness; myths about pain; activity pacing; acceptance and values based goal setting). Patients randomized to this arm gain access to a website downloaded on their phones as an app. The website includes explainer videos of skills and recordings of mindfulness and relaxation exercises. In addition, participants will receive usual care as determined by their medical team.
- Minimally Enhanced Usual Care (MEUC) - Control: In the Minimally Enhanced Usual Care (MEUC) arm of the study, patients who are randomized to this arm will receive educational material, in the form of a physical hard-copy pamphlet and website downloaded as an app on their phones. In addition, these participants will receive usual care as determined by their medical team.
Period: Overall Study
Arm/Group | Toolkit for Optimal Recovery After Orthopedic Injury (TOR) - Active | Minimally Enhanced Usual Care (MEUC) - Control
Started | 97 | 98
Completed | 74 | 81
Not Completed | 23 | 17

BASELINE CHARACTERISTICS:
Population: Participants were individuals with recent orthopaedic injuries (1-2 months prior) with elevator pain anxiety and/or pain catastrophizing.
Groups:
- Toolkit for Optimal Recovery After Orthopedic Injury - Active: Toolkit for Optimal Recovery after Orthopedic Injury: The Toolkit (TOR) is a 4-session, individual, live video, synchronous program developed specifically for patients with orthopedic acute injuries who are at risk for chronic pain and disability. The program teaches evidence-based mind-body skills (e.g., relaxation and mindfulness; myths about pain; activity pacing; acceptance and values based goal setting). Patients randomized to this arm gain access to a website downloaded on their phones as an app. The website includes explainer videos of skills and recordings of mindfulness and relaxation exercises. In addition, participants will receive usual care as determined by their medical team.
- Total: Total of all reporting groups
Arm/Group | Toolkit for Optimal Recovery After Orthopedic Injury - Active | Minimally Enhanced Usual Care (MEUC) - Control | Total
Number analyzed (Participants) | 97 | 98 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (17) | 45 (16) | 44 (17)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Man | 31 | 32 | 63
  Woman | 63 | 62 | 125
  Genderqueer/gender fluid/nonbinary | 3 | 3 | 6
  Prefer not to say | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 66 | 131
  Male | 32 | 32 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 13 | 27
  Not Hispanic or Latino | 80 | 83 | 163
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 76 | 73 | 149
  More than one race | 5 | 7 | 12
  Unknown or Not Reported | 5 | 4 | 9
Education [Count of Participants; unit: Participants]
  Less than high school | 1 | 6 | 7
  Completed high school or GED | 20 | 26 | 46
  Some college/Associates degree | 29 | 23 | 52
  Completed 4 years of college | 30 | 19 | 49
  Graduate/professional degree | 15 | 23 | 38
  Choose Not to Answer | 2 | 1 | 3
Employment [Count of Participants; unit: Participants]
  Employed full-time | 48 | 49 | 97
  Employed part-time | 15 | 9 | 24
  Going to school full or part-time | 4 | 2 | 6
  Keeping House/Housemaker | 1 | 2 | 3
  Other | 3 | 7 | 10
  Retired | 10 | 8 | 18
  Unemployed | 15 | 16 | 31
  Choose Not to Answer | 1 | 5 | 6
Income [Count of Participants; unit: Participants]
  Less than $10,000 | 9 | 17 | 26
  $10,000 to less than $15,000 | 5 | 6 | 11
  $15,000 to less than $20,000 | 4 | 0 | 4
  $20,000 to less than $25,000 | 9 | 3 | 12
  $25,000 to less than $35,000 | 10 | 7 | 17
  $35,000 to less than $50,000 | 14 | 11 | 25
  $50,000 to less than $75,000 | 6 | 12 | 18
  $75,000 or more | 25 | 28 | 53
  Choose Not to Answer | 15 | 14 | 29
Marital Status [Count of Participants; unit: Participants]
  Single, never married | 40 | 36 | 76
  Married | 35 | 39 | 74
  Living with significant other | 4 | 4 | 8
  Separated/Divorced | 12 | 14 | 26
  Widowed | 6 | 4 | 10
  Choose Not to Answer | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Recruitment Among All Patients
Description: We will report number of participants who consented to participate out of those eligible, evaluated at the end of study. This number is not the same as the number who were actually enrolled and randomized in the trial (195).
Time Frame: At the end of the entire enrollment period of the study, which was about 1 year and 10 months.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants (TOR and MEUC): Includes all individuals who were eligible to participate (adult with recent, acute orthopedic trauma) across all four sites.
Arm/Group | All Participants (TOR and MEUC)
Number analyzed (Participants) | 235
Participants | 210

2. Primary Outcome: Appropriateness of Treatment Program, Rated by Participants Randomized to TOR and Assessed by the Credibility and Expectancy Scale
Description: A measure of participant's expectations and believed credibility for program (i.e. appropriateness), as assessed by the Credibility and Expectancy Scale. This scale has a range of 3 to 27 points, with higher ratings indicating more belief that the program is logical and will help with the intended outcome. This measure was the count of patients who scored above or below the scale's theoretical midpoint (i.e. the midpoint is not based on the collected data) on the Credibility and Expectancy Scale
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- TOR Only: Participants who were randomized to TOR after completing baseline assessments. Includes total participants at all four sites (MGH, Dell, VUMC, UK).
Arm/Group | TOR Only
Number analyzed (Participants) | 90
Participants | 66

3. Primary Outcome: Feasibility of Data Collection
Description: This outcome will assess the feasibility of collecting the data used to assess and compare the TOR intervention to MEUC (usual care); it is not looking at the data itself or comparing two arms, but just the feasibility of collecting it. To assess this feasibility marker of our intervention, we will report the number of patients who complete their study assessments, for both TOR and MEUC together, at all of their required timepoints in the study.
Time Frame: On the participant level, data was collected over the course of 4 months (baseline through followup). Counts reported here and described above were summed at the final end of all study activities (a total duration of 1 year 10 months).
Population: Participants in both the active treatment arm (TOR) and control group (MEUC) are reported together, since regardless of study arm, all participants completed the same baseline, posttest, and followup questionnaires at the timepoints. This is appropriate for the feasibility benchmark of data collection; we are only assessing the feasibility of collecting these questionnaires for this outcome across the study as a whole, and not comparing the feasibility between the arms.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants (TOR and MEUC): Includes all individuals who were enrolled across the four sites (MGH, Dell, VUMC, UK).
Arm/Group | All Participants (TOR and MEUC)
Number analyzed (Participants) | 195
Participants | 154

4. Primary Outcome: Acceptability of Treatment (Satisfaction) Assessed With the Client Satisfaction Questionnaire (Patients Randomized to TOR Only)
Description: Participant's satisfaction with treatment received after completion of TOR was assessed using the Client Satisfaction Questionnaire. In this questionnaire, items are summed to generate a total score; scores range from 3 to 12, with higher values indicating higher satisfaction. This measure is the count of participants in TOR who scored above the scale's theoretical midpoint (i.e. the midpoint is not based on the collected data) on the Client Satisfaction Questionnaire.
Time Frame: Assessed at Post-Test, which was approximately 4 weeks after a participant's enrollment in the study and baseline assessment.
Population: The number of participants analyzed in this outcome reflects the number of participants (out of the total enrolled and randomized) who made it to the posttest assessment and could complete this questionnaire (i.e. did not drop out and were not lost to followup in the time since randomization and enrollment).
Measure: Count of Participants; unit: Participants
Arm/Group | TOR Only
Number analyzed (Participants) | 76
Participants | 75

5. Primary Outcome: Acceptability of TOR (Attendance for Patients Randomized to TOR)
Description: We will the report total number of patients in the TOR intervention who attend all four sessions that are part of their intervention.
Time Frame: On the participant level, the data for this outcome was collected over the course of the intervention and its sessions (4 weeks). Counts of attendance were summed at the end of the study (~1 year and 10 months).
Measure: Count of Participants; unit: Participants
Arm/Group | TOR Only
Number analyzed (Participants) | 97
Participants | 71

6. Secondary Outcome: Feasibility of Randomization/Adherence to Assigned Arm, for All Enrolled Patients
Description: We will report number of participants who are randomized within one arm and complete post-test.
Time Frame: Assessed the counts for the study as a whole at the end of study completion, which was about 1 year and 10 months. On the participant level, the time from randomization to posttest took place over an average of 4 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Toolkit for Optimal Recovery After Orthopedic Injury - Active | Minimally Enhanced Usual Care (MEUC) - Control
Number analyzed (Participants) | 97 | 98
Participants | 76 | 93

7. Secondary Outcome: Orthopedic Staff Feasibility of Referral
Description: We will report the number of surgeons and staff who make at least 5 referrals across all four sites, to assess whether referrals for this trial (and thus our intervention) are feasible for surgeons and clinic staff to complete. Referrals could come from providers at any point over the course of the intervention/study.
Time Frame: On the staff member level, the data for this outcome was collected over the course of the entire intervention/study (about 1 year and 7 months total from the start of referrals and participant enrollment in the study).
Population: The active treatment arm (TOR) and control group (MEUC) are not relevant to this outcome/analysis population, since this measure refers to referrals, from surgeons and staff, to the study overall, and it is not related to the actual treatment arms themselves. This is appropriate for the feasibility benchmark assessing whether referrals for this trial (and thus our intervention) are feasible for surgeons and clinic staff to complete.
Measure: Count of Participants; unit: Participants
Groups:
- Referring Staff (All Four Sites Combined): Includes surgeons and staff from all four sites that referred participants and/or facilitated "warm hand-offs" to aid in recruitment.
Arm/Group | Referring Staff (All Four Sites Combined)
Number analyzed (Participants) | 28
Participants | 25

8. Secondary Outcome: Fidelity to Study Procedures (Minor Deviations)
Description: We will report number of minor deviations per each separate, site among all enrolled patients (both TOR and MEUC combined at each site). This is appropriate for the fidelity benchmark of collecting minor deviations; we are only assessing our ability to adhere to the study procedures consistently and not drift in administration (i.e. fidelity), and we are not comparing fidelity in any way between the arms.
Time Frame: On the participant level, the data for this outcome was collected over the course of the intervention as well as the through the followup time point, a total of 4 months. Counts of deviations were summed at the end of the study (~1 year and 10 months).
Population: Total number of participants enrolled per site listed here. Deviations reported for each site are for TOR and MEUC together, since regardless of study arm, deviations were reported and logged for all arms together at each site. This is appropriate for the fidelity benchmark of collecting minor deviations; we are only assessing our ability to adhere to the study procedures consistently and not drift in administration (i.e. fidelity), and we are not comparing fidelity in any way between the arms.
Measure: Number; unit: minor protocol deviations
Groups:
- Massachusetts General Hospital: Team at the Center for Health Outcomes and Interdisciplinary Research at Massachusetts General Hospital
- Dell Medical School: Department of Surgery and Perioperative Care, Dell Medical School
- Vanderbilt University Medical Center: Department of Physical Medicine & Rehabilitation, Osher Center for Integrative Health, Vanderbilt University Medical Center
- University of Kentucky College of Medicine: Department of Orthopaedic Surgery & Sports Medicine, University of Kentucky College of Medicine
Arm/Group | Massachusetts General Hospital | Dell Medical School | Vanderbilt University Medical Center | University of Kentucky College of Medicine
Number analyzed (Participants) | 66 | 48 | 30 | 51
minor protocol deviations | 7 | 1 | 4 | 3

9. Secondary Outcome: Fidelity to Study Procedures (Major Deviations)
Description: We will report number of major deviations per each separate site among all enrolled patients (both TOR and MEUC combined at each site). This is appropriate for the fidelity benchmark of collecting major deviations; we are only assessing our ability to adhere to the study procedures consistently and not drift in administration (i.e. fidelity), and we are not comparing fidelity in any way between the arms.
Time Frame: as for outcome 8
Population: Total number of participants enrolled per site listed here. Deviations reported for each site are for TOR and MEUC together, since regardless of study arm, deviations were reported and logged for all arms together at each site. This is appropriate for the fidelity benchmark of collecting major deviations; we are only assessing our ability to adhere to the study procedures consistently and not drift in administration (i.e. fidelity), and we are not comparing fidelity in any way between the arms.
Measure: Number; unit: major protocol deviations
Arm/Group | Massachusetts General Hospital | Dell Medical School | Vanderbilt University Medical Center | University of Kentucky College of Medicine
Number analyzed (Participants) | 66 | 48 | 30 | 51
major protocol deviations | 1 | 0 | 0 | 0

10. Secondary Outcome: Adherence to TOR Homework
Description: The number of participants who returned at least 1 out of 3 homework logs (1 log was given per week), that have 4 out of 7 days of practice reported on those logs.
Time Frame: On the participant level, the data for this outcome was collected over the course of the intervention and its sessions (4 weeks). Counts were then summed at the end of the study (~1 year and 10 months).
Measure: Count of Participants; unit: Participants
Arm/Group | TOR Only
Number analyzed (Participants) | 97
Participants | 74

11. Secondary Outcome: Acceptability as Rated by Therapist
Description: Assessed using a therapist scale rating patient participation quality in each session. We will report the number of TOR sessions that scored over 7 (out of 10 possible points). There were 304 total TOR sessions delivered over the course of the study, and 294 sessions received a score over 7.
Time Frame: On the participant level, the data for this outcome was collected over the course of the intervention and its sessions (4 weeks). Counts that met our criteria noted in the description were then summed at the end of the study (~1 year and 10 months).
Population: This measure refers to the total number of sessions that were analyzed for this outcome. The overall number of units analyzed that is reported here reflects the total number of sessions delivered over the course of the study, that were then scored by therapists. The overall number of participants analyzed is the number of participants who were randomized to the TOR arm of the study, and received the intervention (which included the sessions (units) that were analyzed for this outcome).
Measure: Number; unit: count of sessions
Units Other Than Participants: Sessions
Groups:
- Fidelity Check - TOR Sessions: Number of sessions in which clinician rated the session > 7 on fidelity checklists
Arm/Group | Fidelity Check - TOR Sessions
Number analyzed (Participants) | 97
Number analyzed (Sessions) | 304
count of sessions | 294

12. Secondary Outcome: Perceived Satisfaction of Staff
Description: We will report the number of surgeons and staff who score over 7 on the satisfaction question that was part of a study feedback survey.
Time Frame: On the staff member level, the data for this outcome was collected in a one-time survey at the end of the intervention and recruitment in their clinics, administered at about 1 year and 7 months from the start of the study.
Population: This population is orthopedic surgeons and staff who were involved with referring patients to the study. The active treatment arm (TOR) and control group (MEUC) are not relevant to this outcome/analysis population, since this measure refers to the satisfaction of surgeons and staff, in regards to the intervention and the study procedures as a whole, and it is not related to the actual treatment arms themselves.
Measure: Count of Participants; unit: Participants
Groups:
- Staff Rating: Includes staff (e.g., surgeons, medical assistants, nurse practitioners, residents) across all four sites that completed a survey after the completion of recruitment to assess staff feasibility and acceptability of the study procedures
Arm/Group | Staff Rating
Number analyzed (Participants) | 20
Participants | 15

13. Secondary Outcome: Perceived Acceptability of Staff Regarding Ease of Referral
Description: We will report number of surgeons and staff who score over 7 on the ease of referral question that was part of a study feedback survey.
Time Frame: as for outcome 12
Population: This population is orthopedic surgeons and staff who were involved with referring patients to the study. The active treatment arm (TOR) and control group (MEUC) are not relevant to this outcome/analysis population, since this measure refers to the perceived acceptability of surgeons and staff, in regards to the intervention and the study procedures as a whole (referral process), and it is not related to the actual treatment arms themselves.
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Rating
Number analyzed (Participants) | 22
Participants | 22

14. Secondary Outcome: Perceived Acceptability of Staff Regarding Cost-benefit for the Patient
Description: We will report the number of surgeons and staff who score over 7 on the cost-benefit (patient) question that was part of a study feedback survey.
Time Frame: as for outcome 12
Population: This population is orthopedic surgeons and staff who referred patients to the study. The active treatment arm (TOR) and control group (MEUC) are not relevant to this outcome/analysis population, since this measure refers to the perceived acceptability of surgeons and staff, in regards to the intervention and cost-benefit to the patient, and it is not related to the actual treatment arms themselves.
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Rating
Number analyzed (Participants) | 19
Participants | 15

15. Secondary Outcome: Perceived Acceptability of Staff Regarding Cost-benefit for the Clinic
Description: We will report the number of surgeons and staff who score over 7 on the cost-benefit (clinic) question that was part of a study feedback survey.
Time Frame: as for outcome 12
Population: This population is orthopedic surgeons and staff who referred patients to the study. The active treatment arm (TOR) and control group (MEUC) are not relevant to this outcome/analysis population, since this measure refers to the acceptability of surgeons and staff, in regards to the intervention and the study procedures (cost-benefit to the clinic) as a whole, and it is not related to the actual treatment arms themselves.
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Rating
Number analyzed (Participants) | 21
Participants | 15

16. Secondary Outcome: Feasibility of Study Implementation as Perceived by Study Staff
Description: We will report the number of surgeons and staff who score over 7 on the feasibility of study implementation question that was part of a study feedback survey.
Time Frame: as for outcome 12
Population: This population is orthopedic surgeons and staff who referred patients to the study. The active treatment arm (TOR) and control group (MEUC) are not relevant to this outcome/analysis population, since this measure refers to the feasibility of implementing the study, as perceived by surgeons and staff, in regards to the intervention and the study procedures as a whole; it is not related to the actual treatment arms themselves.
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Rating
Number analyzed (Participants) | 19
Participants | 15

17. Secondary Outcome: Appropriateness as Perceived by Study Staff
Description: We will report the number of surgeons and staff who score over 7 on the appropriateness question that was part of a study feedback survey. This question assessed the the perceived appropriateness (relevance, compatibility) of the study for their patient population.
Time Frame: as for outcome 12
Population: This population is orthopedic surgeons and staff who referred patients to the study. The active treatment arm (TOR) and control group (MEUC) are not relevant to this outcome/analysis population, since this measure refers to the perceived appropriateness (relevance, compatibility) of the study for their patient population, in regards to the intervention and the study procedures as a whole; it is not related to the actual treatment arms themselves.
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Rating
Number analyzed (Participants) | 16
Participants | 14

18. Secondary Outcome: Feasibility of Obtaining Data on Orthopedic Staff Satisfaction
Description: We will report the number of surgeons and study staff who complete the study feedback survey.
Time Frame: as for outcome 12
Population: This population is orthopedic surgeons and staff who referred patients to the study. The active treatment arm (TOR) and control group (MEUC) are not relevant to this outcome/analysis population, since this measure refers to the feasibility of obtaining the data on staff satisfaction, in regards to the intervention and the study procedures as a whole; it is not related to the actual treatment arms themselves.
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Rating
Number analyzed (Participants) | 22
Participants | 20

19. Secondary Outcome: Feasibility of Obtaining Data on Orthopedic Staff Perceived Ease of Referrals
Description: We will report the number of surgeons and staff who complete the ease of referral question that was part of a study feedback survey.
Time Frame: as for outcome 12
Population: This population is orthopedic surgeons and staff who referred patients to the study. The active treatment arm (TOR) and control group (MEUC) are not relevant to this outcome/analysis population, since this measure refers to the feasibility of obtaining the data on staff ease of referrals, in regards to the intervention and the study procedures as a whole; it is not related to the actual treatment arms themselves.
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Rating
Number analyzed (Participants) | 22
Participants | 22

20. Secondary Outcome: Feasibility of Obtaining Data on Orthopedic Staff Perceived Cost-benefit (Patient) Measure
Description: We will report the number of surgeons and staff who complete the perceived cost-benefit (patient) measure question that was part of a study feedback survey.
Time Frame: as for outcome 12
Population: This population is orthopedic surgeons and staff who referred patients to the study. The active treatment arm (TOR) and control group (MEUC) are not relevant to this outcome/analysis population, since this measure refers to the feasibility of obtaining the data on staff perceived cost-benefit measure for the patient. This is in regards to the intervention and the study procedures as a whole, and is not related to the actual treatment arms themselves.
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Rating
Number analyzed (Participants) | 22
Participants | 19

21. Secondary Outcome: Feasibility of Obtaining Data on Orthopedic Staff Perceived Cost-benefit (Clinic) Measure
Description: We will report the number of surgeons and staff who complete the perceived cost-benefit (clinic) measure question that was part of a study feedback survey.
Time Frame: as for outcome 12
Population: This population is orthopedic surgeons and staff who referred patients to the study. The active treatment arm (TOR) and control group (MEUC) are not relevant to this outcome/analysis population, since this measure refers to the feasibility of obtaining the data on staff perceived cost-benefit measure for the clinic. This is in regards to the intervention and the study procedures as a whole, and is not related to the actual treatment arms themselves.
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Rating
Number analyzed (Participants) | 22
Participants | 21

22. Secondary Outcome: Feasibility of Obtaining Data on Orthopedic Staff Feasibility of Study Implementation
Description: We will report the number of surgeons and staff who complete the feasibility question that was part of a study feedback survey.
Time Frame: as for outcome 12
Population: This population is orthopedic surgeons and staff who referred patients to the study. The active treatment arm (TOR) and control group (MEUC) are not relevant to this outcome/analysis population, since this measure refers to the feasibility of obtaining the data on staff feasibility of study implementation in their clinic. This is in regards to the intervention and the study procedures as a whole, and is not related to the actual treatment arms themselves
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Rating
Number analyzed (Participants) | 22
Participants | 19

23. Secondary Outcome: Feasibility of Obtaining Data on Orthopedic Staff Perceived Appropriateness
Description: We will report the number of surgeons and staff who complete the perceived appropriateness measure question that was part of a study feedback survey.
Time Frame: as for outcome 12
Population: This population is orthopedic surgeons and staff who referred patients to the study. The active treatment arm (TOR) and control group (MEUC) are not relevant to this outcome/analysis population, since this measure refers to the feasibility of obtaining the data on staff perceived appropriateness. This is in regards to the intervention and the study procedures as a whole, and is not related to the actual treatment arms themselves.
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Rating
Number analyzed (Participants) | 22
Participants | 16

24. Secondary Outcome: Numerical Rating Scale (Pain at Rest), Change Between Time Points
Description: Rating of participant's pain at rest using the Numerical Rating Scale, a Likert scale with 0 being no pain and 10 being the worst possible pain. Means reported reflect the Mean Difference between the timepoints noted in the row title.
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-up (3 Months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Toolkit for Optimal Recovery After Orthopedic Injury - Active | Minimally Enhanced Usual Care (MEUC) - Control
Number analyzed (Participants) | 97 | 98
score on a scale
  Baseline to Post-Treatment | -1.7 [-2.1 to -1.2] | -0.5 [-0.9 to -0.1]
  Baseline to Follow-Up | -2.0 [-2.5 to -1.5] | -1.0 [-1.5 to -0.5]

25. Secondary Outcome: Numerical Rating Scale (Pain During Activity), Change Between Time Points
Description: Rate of participant's pain with activity using the Numerical Rating Scale, a Likert scale with 0 being no pain and 10 being the worst possible pain. Means reported reflect the Mean Difference between the timepoints noted in the row title.
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-up (3 Months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Toolkit for Optimal Recovery After Orthopedic Injury - Active | Minimally Enhanced Usual Care (MEUC) - Control
Number analyzed (Participants) | 97 | 98
score on a scale
  Baseline to Post-Treatment | -1.7 [-2.1 to -1.2] | -1.0 [-1.4 to -0.6]
  Baseline to Follow-Up | -2.4 [-3.0 to -1.8] | -1.6 [-2.1 to -1.0]

26. Secondary Outcome: Short Musculoskeletal Function Assessment (SMFA), Change Between Time Points
Description: The Short Musculoskeletal Function Assessment (SMFA) assesses one's self-report physical function and the extent to which a participant is bothered by their functioning. Scores range from 46 to 230. Higher scores represent greater dysfunction or bother. Means reported reflect the Mean Difference between the time points noted in the row title. A decrease in score between baseline and posttest or baseline and followup (i.e. a more negative difference, or larger negative difference, as reported here) reflects improvements in physical function.
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-up (3 Months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Toolkit for Optimal Recovery After Orthopedic Injury - Active | Minimally Enhanced Usual Care (MEUC) - Control
Number analyzed (Participants) | 97 | 98
score on a scale
  Posttest minus baseline mean score | -16 [-19 to -13] | -8 [-11 to -6]
  Followup minus baseline mean score | -24 [-27 to -20] | -18 [-21 to -14]

27. Secondary Outcome: Center for Epidemiologic Study of Depression (CES-D), Change Between Time Points
Description: The Center for Epidemiologic Study of Depression (CES-D), a 20-item measure assesses depressive symptomatology; scores range from 0-60 and higher scores indicate greater depressive symptomatology. Means reported reflect the Mean Difference between the timepoints noted in the row title.
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-up (3 Months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Toolkit for Optimal Recovery After Orthopedic Injury - Active | Minimally Enhanced Usual Care (MEUC) - Control
Number analyzed (Participants) | 97 | 98
score on a scale
  Baseline to post-test | -9 [-11 to -7] | -3 [-5 to -1]
  Baseline to follow-up | -10 [-12 to -7] | -4 [-7 to -2]

28. Secondary Outcome: PTSD Checklist- Civilian Measure (PCL-C), Change Between Time Points
Description: The 17-item PTSD Checklist civilian measure assesses post-traumatic stress; scores range from 17-85 with higher scores indicating greater post-traumatic stress. Means reported reflect the Mean Difference between the timepoints noted in the row title.
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-up (3 Months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Toolkit for Optimal Recovery After Orthopedic Injury - Active | Minimally Enhanced Usual Care (MEUC) - Control
Number analyzed (Participants) | 97 | 98
score on a scale
  Baseline to post-test | -7 [-10 to -5] | -4 [-6 to -1]
  Baseline to follow-up | -10 [-13 to -7] | -5 [-8 to -2]

29. Secondary Outcome: Pain Catastrophizing Scale (PCS), Change Between Time Points.
Description: The Pain Catastrophizing Scale (PCS), a 13-item measure assesses hopelessness, helplessness and rumination about pain, with items ranging from 0-4 and total scores ranging from 0-52, with higher scores indicating higher levels of pain catastrophizing. Means reported reflect the Mean Difference between the timepoints noted in the row title.
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-up (3 Months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Toolkit for Optimal Recovery After Orthopedic Injury - Active | Minimally Enhanced Usual Care (MEUC) - Control
Number analyzed (Participants) | 97 | 98
score on a scale
  Baseline to post-test | -14 [-16 to -12] | -6 [-8 to -4]
  Baseline to follow-up | -15 [-18 to -12] | -8 [-10 to -5]

30. Secondary Outcome: Pain Anxiety Scale, Short Form (PASS-20), Change Between Time Points
Description: The Pain Anxiety Scale, short form (PASS-20) assesses cognitive and somatic symptoms of anxiety, items range from 0-100 and higher scores indicating greater pain anxiety. Means reported reflect the Mean Difference between the timepoints noted in the row title.
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-up (3 Months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Toolkit for Optimal Recovery After Orthopedic Injury - Active | Minimally Enhanced Usual Care (MEUC) - Control
Number analyzed (Participants) | 97 | 98
score on a scale
  Baseline to post-test | -38 [-41 to -34] | -13 [-17 to -10]
  Baseline to follow-up | -38 [-42 to -33] | -19 [-23 to -14]

31. Secondary Outcome: Measure of Current Status (MOCS-A), Change Between Time Points.
Description: The Measure of Current Status (MOCS-A) assesses ability to engage in healthy coping skills, with items ranging from 0-4, total score ranging from 0-52, and higher scores reflect greater self-perceived current state. Means reported reflect the Mean Difference between the timepoints noted in the row title.
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-up (3 Months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Toolkit for Optimal Recovery After Orthopedic Injury - Active | Minimally Enhanced Usual Care (MEUC) - Control
Number analyzed (Participants) | 97 | 98
score on a scale
  Baseline to post-test | 0.4 [0.2 to 0.5] | 0.01 [-0.1 to 0.2]
  Baseline to follow-up | 0.4 [0.3 to 0.6] | 0.1 [-0.03 to 0.3]

32. Secondary Outcome: Cognitive and Affective Mindfulness Scale- Revised (CAMS-R), Change Between Time Points.
Description: The Measure of Current Status (MOCS-A) assesses mindfulness, with total score ranging from 12-48. Higher scores indicate greater mindfulness. Means reported reflect the Mean Difference between the timepoints noted in the row title.
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-up (3 Months)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Toolkit for Optimal Recovery After Orthopedic Injury - Active | Minimally Enhanced Usual Care (MEUC) - Control
Number analyzed (Participants) | 97 | 98
score on a scale
  Baseline to post-test | 3 [2 to 4] | 0 [-1 to 1]
  Baseline to follow-up | 3 [1 to 4] | 1 [-1 to 2]

33. Secondary Outcome: Feasibility of Data Collection of Rescue Analgesics (Non-narcotic)
Description: We will report number of participants with complete data on non-narcotic rescue analgesics (non-narcotic) among all enrolled patients with orthopedic injuries, via self-report log. This is appropriate for the feasibility benchmark of collecting non-narcotic rescue analgesics; we are only assessing our ability to feasibly collect this information, and we are not comparing feasibility in any way between the arms.
Time Frame: On the participant level, the data for this outcome was collected over the course of the intervention as well as the through the followup time point, a total of 4 months. Counts of complete data were summed at the end of the study (~1 year and 10 months).
Population: The data reported are for TOR and MEUC together, since regardless of study arm, any use of non-narcotic rescue analgesics were reported and logged for all arms together. This is appropriate for the feasibility benchmark of collecting non-narcotic rescue analgesics; we are only assessing our ability to feasibly collect this information, and we are not comparing feasibility in any way between the arms.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants (TOR and MEUC)
Number analyzed (Participants) | 195
Participants | 155

34. Secondary Outcome: Feasibility of Data Collection of Rescue Analgesics (Narcotic)
Description: We will report number of participants with complete data on narcotic rescue analgesics among all enrolled patients with orthopedic injuries, via self-report log. This is appropriate for the feasibility benchmark of collecting narcotic rescue analgesics; we are only assessing our ability to feasibly collect this information, and we are not comparing feasibility in any way between the arms.
Time Frame: as for outcome 33
Population: The data reported are for TOR and MEUC together, since regardless of study arm, any use of narcotic rescue analgesics were reported and logged for all arms together. This is appropriate for the feasibility benchmark of collecting narcotic rescue analgesics; we are only assessing our ability to feasibly collect this information, and we are not comparing feasibility in any way between the arms.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants (TOR and MEUC)
Number analyzed (Participants) | 195
Participants | 155

35. Secondary Outcome: Adverse Events (Serious and Non-serious)
Description: We will report number of adverse events (serious and non-serious) per each separate site among all enrolled patients with orthopedic injuries (both TOR and MEUC combined at each site). This is appropriate to report the arms together because we are not comparing adverse events in any way between the arms.
  Definition of an adverse event in this study: throughout the study, subjects were monitored for the occurrence of events defined as any undesirable experience or unanticipated risk. Lack of effect of treatment was not considered an event.
Time Frame: as for outcome 33
Population: Total number of participants enrolled per site are listed here. The adverse events reported below for each site are for TOR and MEUC together, since regardless of study arm, adverse events were reported and logged for all arms together at each site. This is appropriate because we are not comparing adverse events in any way between the arms.
Measure: Number; unit: adverse events
Arm/Group | Massachusetts General Hospital | Dell Medical School | Vanderbilt University Medical Center | University of Kentucky College of Medicine
Number analyzed (Participants) | 66 | 48 | 30 | 51
adverse events
  Adverse Events | 0 | 2 | 0 | 1
  Serious Adverse Events | 1 | 0 | 1 | 1

36. Secondary Outcome: Feasibility of Data Collection of Adverse Events
Description: We will report number of participants with completed data on their adverse events, among enrolled patients with orthopedic injuries in the TOR arm. Data will be reported by study clinicians, for all sites and both arms combined. This is appropriate for the feasibility benchmark of collecting the adverse event data, since we are interested in whether it is feasible for our treatment/study intervention, which is part of the TOR arm only.
Time Frame: On the participant level, data for this outcome was collected over the course of the intervention as well as the through the followup time point, a total of 4 months. Counts of complete data were summed at the end of the study (~1 year and 10 months).
Population: The total number of participants randomized in the TOR arm is listed here. The completed data on adverse events reported below is only for TOR. This is appropriate for the feasibility benchmark of collecting the adverse event data, since we are interested in whether it is feasible for our treatment, which is part of the TOR arm only.
Measure: Number; unit: participants with completed data
Arm/Group | TOR Only
Number analyzed (Participants) | 97
participants with completed data | 97

37. Secondary Outcome: Therapist Adherence/Fidelity to Session
Description: We will report the number of adherence/fidelity "points" that therapists achieved from reviewers during their fidelity checks, over the course of the study. These fidelity checks were done by assessing a checklist review of audio recordings of the sessions, and were completed by 2 raters, for 16 different TOR therapists.
Time Frame: On the fidelity reviewer level, the data for this outcome was collected over the course of the intervention as the sessions were delivered by therapists (4 weeks of delivery). Reviews/points were then summed at end of the study (~1 year and 10 months).
Population: 16 clinicians/therapists were randomly selected to review fidelity checks. Since study clinicians were only used in the intervention arm (TOR), study arm, i.e. TOR vs. MEUC, is not an applicable breakdown for this outcome, as those in the MEUC arm would not have received the intervention, i.e. the sessions that were assessed in this fidelity check.
Measure: Count of Units; unit: Points
Units Other Than Participants: Points
Groups:
- Fidelity Check: TOR Clinicians who were assessed in this fidelity check/outcome
Arm/Group | Fidelity Check
Number analyzed (Participants) | 16
Number analyzed (Points) | 7360
Points | 6829

38. Secondary Outcome: Within-group Use of Rescue Analgesics (Non-narcotic)
Description: Self-report of past-week rescue analgesics use was collected from participants at each assessment timepoint and is reported here for each timepoint; timepoint is indicated in the row title.
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-up (3 Months)
Population: The overall number of participants analyzed reflects all participants who were analyzed at the first timepoint/row below (i.e. baseline). The actual numbers analyzed, reported at each timepoint/row below, reflects that some were lost to follow-up or had dropped out of the study by the different time points.
Measure: Number; unit: percentage
Arm/Group | Toolkit for Optimal Recovery After Orthopedic Injury - Active | Minimally Enhanced Usual Care (MEUC) - Control
Number analyzed (Participants) | 83 | 98
percentage
  Baseline non-narcotic use (percentage) | 22.9 | 64.3
  Post-test non-narcotic use (percentage): number analyzed (Participants) | 76 | 94
  Post-test non-narcotic use (percentage) | 9.2 | 60.6
  Follow-up non-narcotic use (percentage): number analyzed (Participants) | 74 | 80
  Follow-up non-narcotic use (percentage) | 9.5 | 61.3

39. Secondary Outcome: Within Group Use of Rescue Analgesics (Narcotic)
Description: as for outcome 38
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-up (3 Months)
Population: as for outcome 38
Measure: Number; unit: percentage
Arm/Group | Toolkit for Optimal Recovery After Orthopedic Injury - Active | Minimally Enhanced Usual Care (MEUC) - Control
Number analyzed (Participants) | 83 | 98
percentage
  Baseline narcotic use (percentage) | 22.9 | 33.7
  Post-test narcotic use (percentage): number analyzed (Participants) | 76 | 94
  Post-test narcotic use (percentage) | 9.2 | 19.1
  Follow-up narcotic use (percentage): number analyzed (Participants) | 74 | 80
  Follow-up narcotic use (percentage) | 9.5 | 13.8

40. Secondary Outcome: 2-tailed Pearson Correlation (TOR and MEUC)
Description: We assessed the correlation between change scores in the Short Musculoskeletal Function Assessment (SMFA) and change scores on the following mechanistic targets of the TOR intervention: Center for Epidemiologic Study of Depression (CES-D), Posttraumatic Stress Disorder Checklist (PCL), Pain Catastrophizing Scale (PCS), Pain Anxiety Scale Short Form (PASS), Measures of Current Status (MOCS), and Cognitive and Affective Mindfulness Scale-Revised (CAMS-R). Change scores reflected the difference in score between baseline (week 0) and post-test (week 4). Possible correlations range from 0-1; the closer a correlation score is to 1, the more correlated (associated, related) the two measures being compared are. This means that the closer a correlation in change scores is to 1, the more related a change in SMFA is to a change in the named mechanistic target of the intervention.
Time Frame: Baseline (Week 0), Post-Test (Week 4)
Measure: Number (95% Confidence Interval); unit: 2-tailed Pearson Correlation (r)
Groups:
- TOR - Active Treatment Group: Participants who were randomized to TOR after completing baseline assessments. Includes total participants at all four sites (MGH, Dell, VUMC, UK).
- MEUC - Control Group: Participants who were randomized to MEUC after completing baseline assessments. Includes total participants at all four sites (MGH, Dell, VUMC, UK).
Arm/Group | TOR - Active Treatment Group | MEUC - Control Group
Number analyzed (Participants) | 97 | 98
2-tailed Pearson Correlation (r)
  SMFA Change-CES-D Change-Correlation | 0.6 [0.428 to 0.724] | 0.7 [0.539 to 0.769]
  SMFA Change-PCL Change Correlation | 0.4 [0.244 to 0.609] | 0.5 [0.364 to 0.662]
  SMFA Change-PCS Change Correlation | 0.3 [0.044 to 0.465] | 0.4 [0.208 to 0.553]
  SMFA Change-PASS Change Correlation | 0.3 [0.072 to 0.486] | 0.5 [0.313 to 0.626]
  SMFA Change-MOCS Change Correlation | -0.2 [-0.407 to 0.027] | -0.3 [-0.473 to -0.098]
  SMFA Change-CAMS-R Change Correlation | -0.2 [-0.389 to 0.049] | -0.3 [-0.489 to -0.118]

41. Secondary Outcome: Physical Function Self-report, Change Between Time Points
Description: The PROMIS Physical Function (v1.0 8b) assesses one's ability to carry out activities that require physical actions, ranging from self-care to social activities to work. Raw scores are converted to T scores, which are standardized scores based on the average in the population (a score of 50 would indicate matching the average score in the reference, general population. T scores range from 8-40, with a higher score reflecting greater physical function and ability to carry out the activity. Means reported reflect the Mean Difference between the time points in the row titles listed. For the differences reported, a bigger difference thus reflects a greater improvement in physical function.
Time Frame: Baseline (0 Weeks), Post-Test (4 Weeks), Follow-up (3 Months)
Measure: Mean (95% Confidence Interval); unit: T score
Arm/Group | Toolkit for Optimal Recovery After Orthopedic Injury - Active | Minimally Enhanced Usual Care (MEUC) - Control
Number analyzed (Participants) | 97 | 98
T score
  Baseline to Post-Treatment | 6 [5 to 8] | 4 [3 to 6]
  Baseline to Follow-Up | 12 [10 to 14] | 11 [9 to 12]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participant, if needed, over the duration of their time in the study (baseline/enrollment through followup, over a 3 month time period).
Description: Participants in both the active treatment arm (TOR) and control group (MEUC) are reported together (although broken down by site), since adverse events were collected as a whole for both TOR and MEUC together.
Arm/Group | Massachusetts General Hospital | Dell Medical School | Vanderbilt University Medical Center | University of Kentucky College of Medicine
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/48 | 0/30 | 0/51
Serious Adverse Events (participants affected / at risk) | 1/66 | 0/48 | 1/30 | 1/51
Other Adverse Events (participants affected / at risk) | 0/66 | 2/48 | 0/30 | 1/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Massachusetts General Hospital (N=66) | Dell Medical School (N=48) | Vanderbilt University Medical Center (N=30) | University of Kentucky College of Medicine (N=51)
Suicide attempt and subsequent hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diagnosis of ankle septic arthritis and hospitalization (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Patient presented to the emergency department with left ankle swelling, and diagnosed with left ankle septic arthritis/left calcaneal osteomyelitis. The patient was treated surgically and was recommended discharge to the home setting.
Pneumonia and hospitalization (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Massachusetts General Hospital (N=66) | Dell Medical School (N=48) | Vanderbilt University Medical Center (N=30) | University of Kentucky College of Medicine (N=51)
Increased pain severity with movement (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall onto ankle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
New onset of jaw pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-26): https://cdn.clinicaltrials.gov/large-docs/96/NCT04973696/Prot_SAP_000.pdf